CLINICAL TRIAL: NCT04316572
Title: ImPROving Cross-sectoral Collaboration Between Primary and Psychosocial Care: A Randomised Controlled Superiority Trial to Compare the Effectiveness of a Mental Health Specialist VIDEo Consultations Model Versus Treatment as Usual in Patients With Depression or Anxiety Disorders in Primary Care
Brief Title: Mental Health Specialist Video Consultations for Primary Care Patients
Acronym: PROVIDE-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Markus Haun, Internal Medicine Specialist and Head of the Junior Research Group PROVIDE, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: S-923/2019
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Depression; Anxiety Disorder
Keywords: primary care; mental health; telemedicine; video consultations; effectiveness; health services research
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mental health specialist video consultation (Experimental): The intervention group will receive five video consultations with psychotherapists directly in the GP's practice.
  The consultations will be carried out via the web portal of a certified video service provider (arztkonsultation ak GmbH). The patient will be located in the GP's practice and the psychotherapist in his practice or another suitable room. Patients are scheduled for five sessions of 50 minutes.
  Interventions: Behavioral: mental health specialist video consultation
- treatment as usual by the GP (No Intervention): Routine treatment by the GP, which may or may not include conversations about psychosocial problems and/or referral to specialised services (e.g., inpatient therapy, counseling, self-help).

INTERVENTIONS:
Behavioral: mental health specialist video consultation — The consultations will be based on a psychodynamic understanding with a solution-oriented stance and will follow a manual:
  Session 1: Getting familiar with the telemental health setting, building a working alliance and deepening diagnostics.
  Session 2: Clarification of the task/objective, focus building, motivational interviewing if necessary.
  Session 3-4: Focused brief interventions e.g. psychoeducation, promotion of social resources, activation of health-promoting lifestyles (sleep hygiene, eating diary, relaxation etc.), work on personal problems and, if necessary, initiation of further specialised treatment.
  Session 5: Ending the intervention, stabilisation, subsequent treatment plan and communicating a case summary to the general practitioner
  Arms: mental health specialist video consultation

SUMMARY:
Even in Western health care systems, most people with mental disorders, including those with severe and chronic disorders, are treated solely by their general practitioner (GP). Notably, the accessibility of mental health specialist care is mainly complicated by (a) long waiting times for specialists, (b) long travel distances to specialists, particularly in rural and remote areas, (c) patients' reservations about mental health specialist care (including fear of being stigmatised by seeking such care). To mitigate those barriers, technology-based integrated care models have been proposed. The purpose of this study is to measure the effectiveness of a mental health specialist video consultations model versus treatment as usual in patients with depression or anxiety disorders in primary care. In an individually randomized, prospective, two-arm superiority study with parallel group design, N = 320 patients with anxiety and/or depressive disorder will be recruited in GP practices.

DETAILED DESCRIPTION:
The purpose of this study is to measure the effectiveness of a mental health specialist video consultations model versus treatment as usual in patients with depression or anxiety disorders in primary care. In total, the investigators plan to enrol 320 patients who will be randomly allocated to the experimental condition (mental health specialist video consultations) or the control condition (treatment as usual from their GP) in a 1:1 ratio. General practitioners will recruit patients during their regular clinic hours. If the patient is interested in participation, the patient will receive the informed consent form and the baseline questionnaire from the GP. The practice team will send the patient's contact details to the study team who will screen the patient with respect to the eligibility criteria.

Patients will be randomly allocated to one of the two study conditions (video consultation model vs. treatment-as-usual, TAU) in a 1:1 ratio by central randomisation.

The evaluation of the primary outcome will be performed according to the intention-to-treat principle.

The health economic evaluation will be carried out from the perspective of society. A cost-effectiveness and a cost-utility analysis will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* at least one of the following psychological conditions i) at least moderately severe depression, defined as a PHQ-9 score of 10 or greater with either item one and/or two being endorsed, ii) at least moderately general anxiety disorder, defined as a Generalized Anxiety Disorder (GAD)-7 score of 10 or greater, or iii) exceeding the cut off of 11 points of the combined anxiety and depression score (PHQ-ADS)
* currently no or as yet insufficient treatment (psychotherapy, psychopharmacotherapy, or both) or difficulty with adherence
* capable of giving consent
* written informed consent

Exclusion Criteria:

* substance abuse/dependence that is likely to compromise intervention adherence
* risk of endangerment to others and/or risk of self-endangerment
* need for emergency medical treatment
* acute psychotic symptoms
* severe cognitive impairment or dementia
* significant hearing and/or visual impairment
* pregnancy in the ≥ 2nd Trimester
* prior experience with video consultations as part of the feasibility trial
* insufficient German language proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
The Patient Health Questionnaire Depression and Anxiety Scale (PHQ-ADS) | 6 months after inclusion
  composite measure of depression and anxiety (range: 0-48 Points, higher score indicates more severly depressed/anxious)

SECONDARY OUTCOMES:
The Patient Health Questionnaire Depression and Anxiety Scale (PHQ-ADS) | 12 months after inclusion
  composite measure of depression and anxiety (range: 0-48 Points, higher score indicates more severly depressed/anxious)
The Patient Health Questionnaire (PHQ-9) | 6 months after inclusion, 12 months after inclusion
  depressive symptom severity (range: 0-27 Points, higher score indicates more severly depressed)
Generalized Anxiety Disorder Scale (GAD-7) | 6 months after inclusion, 12 months after inclusion
  anxiety symptom severity, range: 0-21, higher score indicates worse outcome
Short-Form Health Survey 12 (SF-12) | 6 months after inclusion, 12 months after inclusion
  health related quality of life (two dimensions: physical and mental quality of life, ranges: 0-100, higher score indicates higher quality of life
Recovery Assessment Scale (RAS-G) | 6 months after inclusion, 12 months after inclusion
  self-reported mental health recovery, five dimension: 1) Goal and success orientation, 2) No domination by Symptoms, 3) Personal confidence and hope, 4) Reliance on others, 5) Willingness to ask others for help, ranges 1-5, higher score indicates better outcome
Somatic Symptom Disorder-B Criteria Scale (SSD-12) | 6 months after inclusion, 12 months after inclusion
  self-reported somatisation, range: 0-48, higher score indicates worse outcome
Patient Assessment of Chronic Illness Care (PACIC) | 6 months after inclusion, 12 months after inclusion
  patients' satisfaction with the care of their chronic disease, range: 1-5, higher score indicates higher satisfaction
EQ-5D | 6 months after inclusion, 12 months after inclusion
  health related quality of life for health economic Evaluations, 5 dimensions: 1) Mobility, 2) Self-Care, 3) Usual Activities, 4) Pain/Discomfort, 5)Anxiety/Depression
Questionnaire for the Assessment of Medical and non Medical Resource Utilisation in Mental Disorders (FIMPsy) | 6 months after inclusion, 12 months after inclusion
  self reported use of medical and psychosocial services for health-economic evaluation

OTHER OUTCOMES:
Assessment of Negative Effects of Psychotherapy (INEP) | 6 months after inclusion, 12 months after inclusion (not measured at baseline, patients in control condition fill in adapted version)
  unintended/adverse effects of the intervention
Normalisation MeAsure Development questionnaire (NoMAD) | 6 months after inclusion, 12 months after inclusion (measured in GPs and study therapists only)
  measurement of acceptance of newly introduced treatment models, 4 dimensions, range:1-5, lower score indicates greater acceptance of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Haun, MD, MSc, Principal Investigator — Department of General Internal Medicine and Psychosomatics, Heidelberg University
Locations (1):
- Heidelberg University, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, Analytic Code

REFERENCES:
- [Derived] Muller S, Ritter-von Kramer A, Tonnies J, Wildenauer A, Wensing M, Friederich HC, Haun MW. Engaging underrepresented patient groups in specialised treatment - qualitative results from the PROVIDE-C randomised trial on integrated mental health video consultations for depression and anxiety. BMC Public Health. 2025 Nov 6;25(1):3817. doi: 10.1186/s12889-025-25235-1. PMID 41199204
- [Derived] van Eickels D, Henning K, Wensing M, Friederich HC, Haun MW. Psychometric validation of the German version of the somatic symptom disorder - B criteria scale (SSD-12) in a primary care population with depression and anxiety: A COSMIN-guided analysis. Gen Hosp Psychiatry. 2025 Nov-Dec;97:3-10. doi: 10.1016/j.genhosppsych.2025.09.001. Epub 2025 Sep 4. PMID 40939424
- [Derived] Haun MW, Tonnies J, Hartmann M, Wildenauer A, Wensing M, Szecsenyi J, Feisst M, Pohl M, Vomhof M, Icks A, Friederich HC. Model of integrated mental health video consultations for people with depression or anxiety in primary care (PROVIDE-C): assessor masked, multicentre, randomised controlled trial. BMJ. 2024 Sep 25;386:e079921. doi: 10.1136/bmj-2024-079921. PMID 39322237
- [Derived] Haun MW, Tonnies J, Krisam R, Kronsteiner D, Wensing M, Szecsenyi J, Vomhof M, Icks A, Wild B, Hartmann M, Friederich HC. Mental health specialist video consultations versus treatment as usual in patients with depression or anxiety disorders in primary care: study protocol for an individually randomised superiority trial (the PROVIDE-C trial). Trials. 2021 May 5;22(1):327. doi: 10.1186/s13063-021-05289-3. PMID 33952313